CLINICAL TRIAL: NCT06745284
Title: An Active-comparator-controlled, Open-label, Parallel Group Study to Evaluate the Effect of Survodutide on Energy Expenditure and Fatty Acid Oxidation in Subjects With Obesity
Brief Title: A Study to Test Whether Survodutide Improves How the Body Uses Energy and Breaks Down Fat in People With Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0045; U1111-1309-3679 (Registry Identifier: WHO register - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-12-19; First posted 2024-12-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Survodutide arm (Experimental)
  Interventions: Drug: Survodutide
- Semaglutide arm (Active Comparator)
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Survodutide — Survodutide
  Other Names: BI 456906
  Arms: Survodutide arm
Drug: Semaglutide — Semaglutide
  Other Names: Wegovy®
  Arms: Semaglutide arm

SUMMARY:
This study is open to adults between 18 and 65 years of age who have obesity. People can join the study if they have a body mass index (BMI) between 30 and 45 km/m². The purpose of this study is to find out whether a medicine called survodutide improves how the body uses energy and breaks down fat. This study compares survodutide with another medicine called semaglutide. Survodutide is being developed to treat people with obesity.

Semaglutide is already used to treat people with obesity.

Participants are put into 2 groups by chance. One group gets survodutide and the other group gets semaglutide. Participants get survodutide or semaglutide as an injection under the skin once a week. Participants are in the study for 8-10 months depending on how long the treatment is given. During this time, they visit the study site weekly. Some of the visits may also be done at the participant's home instead of the study site.

At some of the visits, doctors test how much energy a participant's body uses. This is done in a special room where they measure the oxygen that is breathed in and the carbon dioxide that is breathed out by the participant. The results are compared between the 2 groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Age of 18 to 65 years (inclusive)
* Male or female subjects with obesity (defined as a body mass index (BMI) of ≥30 and ≤45 kg/m²)
* Woman of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information
* Signed and dated written informed consent in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* In the investigator's opinion, are well-motivated, capable, and willing to:

  * Learn how to self-inject the investigational medicinal product (IMP), as required for this protocol (persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject the IMP)
  * Inject the IMP or accept injection from a designated person --- Follow trial procedures for the duration of the trial, including, but not limited to: follow lifestyle advice (for example, dietary restrictions and exercise, maintain a diary, complete required questionnaires, and handle the IMP as described in the instruction for use (IFU))

Exclusion criteria:

* Current or history of significant alcohol consumption (defined as intake of >210 g/week in men and >140 g/week in women on average over a consecutive period of more than 3 months) or are unwilling to stop alcohol consumption 48 h before admission to the research facility and until discharge
* History of chronic liver disease / cirrhosis
* Body weight variation (self-reported) >5% within 3 months before Visit 1 (screening)
* Medications for obesity (including over-the-counter medications) within 3 months before Visit 1 (screening)
* Glycated haemoglobin (HbA1c) ≥6.5% (≥48 mmol/mol) as measured by the local laboratory at screening
* History of type 1 diabetes mellitus (T1DM) or T2DM or treatment with glucose lowering agent started within 3 months before Visit 1 (screening) Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
Absolute change in sleeping metabolic rate (SMR) (measured in a whole room calorimeter) from baseline to first visit a participant reached at least 10% weight loss | at baseline, up to 36 weeks

SECONDARY OUTCOMES:
Relative change in SMR (measured in a whole room calorimeter) from baseline to first visit a participant reached at least 10% weight loss | at baseline, up to 36 weeks
Absolute change in fatty acid oxidation during sleep (measured in a whole room calorimeter) from baseline to first visit a participant reached at least 10% weight loss | at baseline, up to 36 weeks
Relative change in fatty acid oxidation during sleep (measured in a whole room calorimeter) from baseline to first visit a participant reached at least 10% weight loss | at baseline, up to 36 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Translational Research Institute for Metabolism and Diabetes, Orlando, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com